CLINICAL TRIAL: NCT04650906
Title: A Feasibility Study for Evaluating the Effectiveness of Mindhelper- a National Youth Mental Health Promotion Website
Brief Title: A Feasibility Study for Evaluating the Effectiveness of Mindhelper - a National Youth Mental Health Promotion Website
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Anna Paldam Folker, Head of Research, Associate professor, PhD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TrygFonden ID: 148711
Record Dates: First submitted 2020-10-23; First posted 2020-12-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Mental Health Issue; Young Adult; Feasibility Studies; Randomized Controlled Trial; Internet-Based Intervention; Recruitment
Keywords: Online recruitment; Denmark

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
  Young people will be recruited through Facebook.dk and instragram, and block randomized to either use of Mindhelper (intervention group) or no information on Mindhelper (control group).
  At baseline participants will respond to a questionnaire on sociodemographic characteristics, and validated items related to well-being (primary outcome), psychological distress and daily functioning (secondary outcomes), and intentions and barriers to help-seeking (explorative outcomes). One week later participants will be asked to respond to a similar questionnaire. We will use 1:1 propensity score to increase comparability between the two groups and report the standardized difference on all baseline variables between high- and low-level users to evaluate whether the matching.
Who Masked: Participant
Masking Description: The participants are partly masked. The control group will be masked; however, the intervention group will not be masked. Other parties will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group gets information about the Mindhelper website and the control group does not get information about the Mindhelper website.
  Interventions: Behavioral: Mindhelper - a national youth mental health promotion website
- Control group (No Intervention): The intervention group gets information about the Mindhelper website and the control group does not get information about the Mindhelper website.

INTERVENTIONS:
Behavioral: Mindhelper - a national youth mental health promotion website — Mindhelper is a fully digital youth mental health service reaching out to a large number of young people when and where they need it, with full anonymity. Mindhelper was developed in 2014-2017 by Centre for Telepsychiatry in the Region of Southern Denmark in a partnership with four Danish municipalities. The development of the site was funded by the Danish foundation TrygFonden. The original idea behind the site was inspired by the Australian youth mental health promotion service ReachOut.com. The Mindhelper service was launched in September 2016. From January 2019 Mindhelper received permanent funding through a joint agreement between the five Danish Regions. Mindhelper is Denmark's most comprehensive youth mental health promotion website where young people can seek mental health information, advice, and self-help tools to improve their mental health and well-being. Since it was launched, the site has been very successful in attracting large numbers of visitors.
  Arms: Intervention group

SUMMARY:
The feasibility study will investigate the potential of online recruitment for a randomized trial of the effectiveness of Mindhelper. Recruiting participants for intervention studies is increasingly difficult, as there are many commercials and research projects competing for people's attention. Thus, participation rates in research projects are generally declining. The widespread access to the internet, especially among adolescents, offers a new and attractive alternative strategy to recruit participants for intervention studies.

The feasibility study will inform us whether it is possible to recruit young people with mental health problems who are not familiar with Mindhelper and then randomize them to use or not to use the website (block randomization). Furthermore, it is necessary to know whether it is possible to follow the two groups over time and assess relevant outcomes.

We aim to answer the following questions:

* Is it possible to identify and recruit young persons (15-25 years of age) in need of mental health promotion via social networking sites such as Facebook.dk?
* How quickly is it possible to recruit people for the study through networking sites?
* Is it possible to ensure that the intervention group uses the Mindhelper website (>75%) and minimize the likelihood that the control group uses it (<25%)?
* Is it possible to follow the two groups to obtain information at first follow-up at one week (T2)?

The results will inform the study design of the effectiveness study. If the feasibility study shows (i) that it is possible to recruit and randomize young people with mental health problems within a specified period, (ii) that both groups will follow their randomization into either the intervention or control group, and (iii) that it is possible to follow both groups to obtain follow-up data, then the main study will be conducted as an online recruited randomized effectiveness study (online RCT). If the feasibility study shows that the conditions are not ideal for achieving these goals, we will conduct a longitudinal panel study of Mindhelper users comparing different types of users.

DETAILED DESCRIPTION:
Introduction Up to 25% of young people in Denmark do not enjoy their daily lives; they report increasing levels of stress, loneliness, sleep problems, and symptoms of anxiety and depression. Online mental health promotion has the potential to address some of the mental health needs of young people. However, the evidence-base for the effectiveness of online mental health promotion is still sparse. The Mindhelper Study will evaluate the effectiveness of the most comprehensive online youth mental health promotion website in Denmark; Mindhelper.dk. Mindhelper is targeted at young people in need of mental health promotion. This is a broad group that encompasses three different subgroups of young people; (i) those who need advice on various well-being issues such as dealing with peer-pressure or a broken heart, (ii) those with early signs of mental health problems, and (iii) those who have mental disorders (or other chronic diseases) who need help to promote their mental health and well-being - such as dealing with loneliness, sleep problems, or structuring their everyday life - alongside more specialized treatment.

The Mindhelper website is designed as a first step in a stepped-care approach to organize the mental health system. At the website, young people are provided trusted mental health information and tools to improve their mental health and well-being. The feasibility study described in this document is the first step of the evaluation.

Feasibility study The feasibility study will investigate the potential of online recruitment for a randomized trial of the effectiveness of Mindhelper. Recruiting participants for intervention studies is increasingly difficult, as there are many commercials and research projects competing for people's attention. Thus, participation rates in research projects are generally declining. The widespread access to the internet, especially among adolescents, offers a new and attractive alternative strategy to recruit participants for intervention studies.

While online recruitment may seem feasible and useful for recruiting subpopulations that are normally difficult to include in intervention studies, such as young people with mental health problems, only few studies have been undertaken. Some studies have examined the feasibility of online recruitment among the general population, couples planning pregnancy, patients with urinary incontinence, and people with drug or alcohol dependencies. The lessons learned from these studies are that the costs per participant are lower, compared to offline recruitment methods; that it is possible to reach populations who are otherwise challenging to enroll because they have sensitive health concerns; and that the recruited persons are younger, more highly educated, and have poorer self-rated health and higher self-efficacy than representative samples. Concerns have been raised that internet- based studies may be particularly prone to selection bias. However, a Danish study of reproductive women showed that internet-based cohorts were not more prone to selection bias than other recruitment methods, which has also been shown among smokers recruited by email or online for a smoking cessation trial.

The feasibility study will inform us whether it is possible to recruit young people with mental health problems who are not familiar with Mindhelper and then randomize them to use or not to use the website (block randomization). Furthermore, it is necessary to know whether it is possible to follow the two groups over time and assess relevant outcomes.

Young people will be recruited through Facebook.dk and Instagram. The first phase of the recruitment will target young people that are in need of mental health promotion, therefore adds for the study will be targeted individuals that have liked or are members of sites on Facebook concerning mental health e.g. the initiative against loneliness Ventilen. Further the initial recruitment will target young people living in the area of Odense, as this is where CTP is placed and therefore will ease the collection of web history. If the investigators do not succeed recruiting all participants with this rather narrow strategy, the investigators will further include the area in and around Copenhagen, as web history may as well be collected at CFI. Hereafter, the recruitment strategy will be widened, to guarantee an uptake of 120 participants. The constant inclusion criteria will be young people aged 15-25, Danish speaking, and Danish residency.

The feasibility study investigates the potential of online recruitment through social media for a randomized trial of the effectiveness of Mindhelper.

The investigators aim to answer the following questions:

* Is it possible to identify and recruit young persons (15-25 years of age) via social networking sites such as Facebook.dk?
* How quickly is it possible to recruit people for the study through networking sites?
* Is it possible to ensure that the intervention group uses the Mindhelper website (>75%) and minimize the likelihood that the control group uses it (<25%)?
* Is it possible to follow the two groups to obtain information at first follow-up at one week (T2)?

The results will inform the study design of the effectiveness study. If the feasibility study shows (i) that it is possible to recruit and randomize young people with mental health problems within a specified period, (ii) that both groups will follow their randomization into either the intervention or control group, and (iii) that it is possible to follow both groups to obtain follow-up data, then the main study will be conducted as an online recruited randomized effectiveness study (online RCT). If the feasibility study shows that the conditions are not ideal for achieving these goals, the investigators will conduct a longitudinal panel study of Mindhelper users comparing different types of users (see description below).

As this is a feasibility study, a formal sample size calculation will not be performed. The investigators plan to include approximately 120 persons (60 in the intervention group and 60 in the control group), which is slightly higher than the standard number. A subsample of the participants will further be invited to the Centre for Telepsychiatry, Mental Health Services in the Region of Southern Denmark, to let a researcher code their web history related to the participants use of Mindhelper. The researcher may view their web history for the past week, but will only code activity related to Mindhelper, which as well is the only information that will be saved and applied in further analyses. This data will also be used to validate survey responses of use of the website, and asses if self-reported questions on online behavior is a valid measure for actual online behavior. Participant who visit the Centre for Telepsychiatry will be given a gift card for the cinema (200 DKK) in appreciation for their participation in the study. Among participants responding to both surveys, there will be a lottery were a few participants will win a gift for the cinema (200 DKK). Participants that are given gifts, will be informed that tax regulations may apply, and that it is their responsibility to inform SKAT of the gift. The financial compensation for participants is given independent of their responds and web history, which give no reason to believe that the gifts may impact the study in any other way, than to promote participations and full follow-up.

Ethics The design of The Mindhelper Study is guided by the CONSORT Statement and the STROBE guidelines. The study will be conducted in accordance with the Danish Council for Independent Research's ethical guidelines. The study will be registered and approved by the University of Southern Denmark in accordance with the Data Protection Regulation and comply with the General Data Protection Regulation (GDPR) (EU) 2016/679. All participants will receive comprehensive information about the purpose of the project and terms of participation. The participants will be asked to give their written consent to participate in the research. The trial will also be registered by ClinicalTrials.gov which is a database of privately and publicly funded clinical provided by the U.S. National Library of Medicine (https://www.clinicaltrials.gov/). The investigators will publish the results of the feasibility study regardless of the outcome.

The study focuses on mental wellbeing and health promotion, not on mental illness nor psychiatric diagnoses, and thus participants may be enrolled independently of their mental health. Broad scales of mental health will primarily be applied in the survey. When sensitive topics as bullying and self-harm occur, it will be related to participants use of Mindhelper, and participants will never be asked for details in this relation, neither will any of the question be on an individual level. However, if a participant respond that he/she e.g. has experienced bullying, or is lonely, he/she will be encouraged to contact organizations able to support him/her (e.g. Børnetelefonen og Ventilen) and contact information will be provided directly in the survey. Participants are eligible for participation if they are between 15 and 25 years of age. According to Danish law children can give consent based on their maturity and children of the aged of 13 years and above can give consent for use of their personal data. However, participants will be encouraged to talk to their parents or other adults if on doubt of participation.

ELIGIBILITY:
Inclusion Criteria:

* aged 15-25
* Danish speaking
* Danish residency

Exclusion Criteria:

* None

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 560 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Possibility to identify and recruit young persons (15-25 years of age) in need of mental health promotion via social networking sites such as Facebook.dk. | Up to 2 months
  Number of participants between 15-25 years of age in need of mental health promotion recruited via social networking sites such as Facebook.dk.
The timeframe for recruiting people for the study through networking sites | Up to 2 months
  Number of days for recruiting people for the study through networking sites
Possibility to ensure that the intervention group uses the Mindhelper website (>75%) and possibility to minimize the likelihood that the control group uses it (<25%)? | Up to 2 months
  Number of participants between 15-25 years of age assigned to the intervention group that uses Mindhelper and number of participants between 15-25 years of age assigned to the control group that does not use it.
Possibility to follow the two groups to obtain information at first follow-up at one week | Up to 2 months
  Number of participants in the intervention and control group who filled the follow-up questionnaire after one week.

CONTACTS AND LOCATIONS:
Overall Officials: Anna P Folker, Principal Investigator — University of Southern Denmark
Locations (2):
- Denmark (2):
  - National Institute of Public Health (NIPH), University of Southern Denmark, Copenhagen
  - Centre for Telepsychiatry (CTP), Mental Health Services in the Region of Southern Denmark, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffmann SH, Paldam Folker A, Buskbjerg M, Paldam Folker M, Huber Jezek A, Lyngso Svarta D, Nielsen Solvhoj I, Thygesen L. Potential of Online Recruitment Among 15-25-Year Olds: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 May 25;6(5):e35874. doi: 10.2196/35874. PMID 35612877